CLINICAL TRIAL: NCT00113191
Title: A Phase III, Randomized, Double-blind, Multi-center Clinical Trial Comparing the Safety and Efficacy of Veronate® Versus Placebo for the Prevention of Nosocomial Staphylococcal Sepsis in Premature Infants (Birth Weight 500 - 1250 g)
Brief Title: Safety and Efficacy of Veronate® Versus Placebo in Preventing Nosocomial Staphylococcal Sepsis in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IgG-CL-006
Record Dates: First submitted 2005-06-06; First posted 2005-06-07 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Nosocomial Infections; Sepsis; Staphylococcal Infections; Candidemia
Keywords: late onset sepsis; premature infants; staphylococcus; candida; prevention
MeSH Terms: conditions — Cross Infection; Sepsis; Staphylococcal Infections; Candidemia; Premature Birth; Torulopsis | interventions — Veronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Veronate

SUMMARY:
The purpose of this study is to show whether Veronate, a donor-selected staphylococcal human immune globulin intravenous (IGIV), can prevent an infection in the blood caused by staphylococcal bacteria in premature babies weighing between 500 and 1250 grams at birth.

Babies are enrolled between Day of Life 3 and 5. Babies are randomized to either Veronate or placebo (50-50 chance of either). Babies can receive up to 4 doses of the study drug on Study Days 1, 3, 8 and 15 and are followed until Study Day 70 or discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from parent or legal guardian
* Birth weight 500 to 1250 g, inclusive
* Age 3 - 5 days (49 to 120 hours), inclusive
* Expected to require IV access for medical care through day of life 14

Exclusion Criteria:

* Already received or likely to receive prior to first infusion of Study Drug:

  * IGIV or *immune globulin for prevention of Hepatitis B
* Receiving an agent for prevention of staphylococcal catheter related or nosocomial infections (e.g., vancomycin)
* Active sepsis, as defined by one of the following:

  * culture proven early onset sepsis and not clinically stable; or
  * clinical signs of sepsis and pending blood cultures; if the blood cultures are negative after 48 hours and the infant is clinically stable, the infant may be randomized
* Severe congenital anomaly, where the prospects for survival, the medical complications and treatment, would compromise the study related outcome evaluation(s) in the Investigator's opinion
* Diagnosis of congenital immunodeficiency
* Evidence of significant fluid overload or significant volume depletion
* Evidence of abnormal renal function as measured by serum creatinine > 1.6 mg/dL

Ages: 3 Days to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2000
Dates: Start 2004-05; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of Veronate® compared to placebo in preventing nosocomial S. aureus sepsis in premature infants
To assess the safety profile of Veronate® compared to placebo in premature infants as measured by frequencies of adverse events, serious adverse events and morbidities associated with prematurity

SECONDARY OUTCOMES:
To compare the proportions of infants with nosocomial coagulase negative staphylococcus (CoNS) sepsis between premature infants treated with Veronate® versus placebo
To compare the proportions of infants with all nosocomial staphylococcal sepsis between premature infants treated with Veronate® versus placebo
To compare the proportions of infants with nosocomial candidemia between premature infants treated with Veronate® versus placebo
To compare mortality between premature infants treated with Veronate® versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Seth V. Hetherington, MD, Study Director — Inhibitex
Locations (82):
- United States (74):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Anchorage, Alaska
  - Phoenix, Arizona
  - Hayward, California
  - Loma Linda, California
  - Long Beach, California
  - Oakland, California
  - Orange, California
  - Sacramento, California
  - San Francisco, California
  - Santa Clara, California
  - Walnut Creek, California
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Plantation, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Honolulu, Hawaii
  - Evanston, Illinois
  - Park Ridge, Illinois
  - Indianapolis, Indiana
  - South Bend, Indiana
  - Wichita, Kansas
  - Baltimore, Maryland
  - Detroit, Michigan
  - Flint, Michigan
  - Grand Rapids, Michigan
  - Lansing, Michigan
  - Royal Oak, Michigan
  - Duluth, Minnesota
  - Jackson, Mississippi
  - St Louis, Missouri
  - Camden, New Jersey
  - Newark, New Jersey
  - Voorhees Township, New Jersey
  - Albany, New York
  - Manhasset, New York
  - Mineola, New York
  - New Hyde Park, New York
  - Syracuse, New York
  - The Bronx, New York
  - Valhalla, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Youngstown, Ohio
  - Bryn Mawr, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wynnewood, Pennsylvania
  - Providence, Rhode Island
  - Greenville, South Carolina
  - Memphis, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Ogden, Utah
  - Provo, Utah
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Spokane, Washington
  - Morgantown, West Virginia
- Canada (8):
  - New Westminster, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - Kingston, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan

REFERENCES:
- [Derived] DeJonge M, Burchfield D, Bloom B, Duenas M, Walker W, Polak M, Jung E, Millard D, Schelonka R, Eyal F, Morris A, Kapik B, Roberson D, Kesler K, Patti J, Hetherington S. Clinical trial of safety and efficacy of INH-A21 for the prevention of nosocomial staphylococcal bloodstream infection in premature infants. J Pediatr. 2007 Sep;151(3):260-5, 265.e1. doi: 10.1016/j.jpeds.2007.04.060. Epub 2007 Jul 24. PMID 17719934